CLINICAL TRIAL: NCT02158988
Title: Prospective Multicenter Phase III Trial Using CRS With / Without HIPEC After Preoperative Chemotherapy in Patients With Peritoneal Carcinomatosis of Gastric Cancer Incl. Adenocarcinoma of the Esophagogastric Junction
Brief Title: Cytoreductive Surgery (CRS) With/Without HIPEC in Gastric Cancer With Peritoneal Carcinomatosis
Acronym: GASTRIPEC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Cancer Aid (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Beate Rau MBA, Prof., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gastripec I
Record Dates: First submitted 2014-05-04; First posted 2014-06-09 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Malignant Neoplasm of Stomach; Secondary Malignant Neoplasm of Peritoneum; Secondary Malignant Neoplasm of Other and Unspecified Sites
Keywords: Gastric cancer; cancer of the esophagogastric junction; peritoneal carcinomatosis; hyperthermic intraperitoneal chemotherapy; HIPEC
MeSH Terms: conditions — Stomach Neoplasms; Peritoneal Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Intervention Model Description: intraperitoneal (in the abdominal cavity) chemoperfusion with Mitomycin C and Cisplatin
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- without HIPEC (No Intervention): Preoperative chemotherapy 3 cycles, each cycle 21 days. Patients with negative or unknown HER-2 status receive Epirubicin 50 mg/m² infusion (maximum 100mg/d). Oxaliplatin 130 mg/m² infusion (maximum 260 mg/d) and capecitabine oral 625 mg/m² two times a day (maximum 2500 mg/d).
  Patients with positive HER-2 status receive:
  Cisplatin : 80 mg/m² infusion (maximum of 160 mg/d). Capecitabine: oral 1000 mg/m2 (two times a day maximum of 4000 mg/d), on day 1-14.
  Trastuzumab: 8 mg/kg infusion (on cycle 1 and 6 mg/kg on cycle 2 and 3). CRS is performed and 4-12 weeks after CRS 3 cycles of postoperative chemotherapy have to be applied. In case of therapy failure patients will be continued to be treated by the responsible investigator according to his medical status.
- With HIPEC (Experimental): Patients will be treated with a preoperative chemotherapy as described for the control group. EOX or CCT depending on the HER-2 status.
  CRS will be performed 2 to 3 weeks after end of last chemotherapy cycle. HIPEC with mitomycin C and cisplatin either at the time of CRS or a delayed HIPEC within 5-7 days.
  HIPEC:
  Mitomycin C: 15 mg/m2 (max. 30 mg/ m2, max. 5 L Perfusion). Cisplatin: 75 mg/m2/L (max. 150 mg/m2, max. 5 L Perfusion). 4-12 weeks after cytoreductive surgery 3 cycles postoperative chemotherapy will be applied.
  Patients may get a HIPEC intervention without surgical cytoreduction if contraindication to the drugs can be excluded.
  In case of therapy failure patients will be continued to be treated by the responsible investigator according to his medical status.
  Interventions: Procedure: HIPEC

INTERVENTIONS:
Procedure: HIPEC — HIPEC:
  Mitomycin C: 15 mg/m2 (max. 30 mg/ m2, max. 5 L Perfusion). Cisplatin: 75 mg/m2/L (max. 150 mg/m2, max. 5 L Perfusion). 4-12 weeks after cytoreductive surgery 3 cycles postoperative chemotherapy will be applied.
  Arms: With HIPEC

SUMMARY:
Patients with histological proven gastric cancer (including cancer of the esophagogastric junction (AEG)) and synchronous peritoneal carcinomatosis, who fulfill the inclusion and exclusion criteria, can be recruited in this study. There are two treatment groups (A and B). The chemotherapy applied intravenously is the same in both groups and is approved for the treatment of gastric cancer. Patients with negative or unknown HER-2 status will be administered Epirubicin, Oxaliplatin and Capecitabine (EOX). Patients with positive HER-2 status will be treated with Cisplatin, Capecitabine and Trastuzumab (CCT).

The chemotherapy is followed by surgical cytoreduction in both groups. Patients randomized into group B will be treated with an intraperitoneal (in the abdominal cavity) chemoperfusion with Mitomycin C and Cisplatin .

Patients in both groups receive 3 cycles of postoperative chemotherapy within 4-12 weeks after the surgical procedure and are followed up for 30 months.

If progress of the tumor is detected the patient will no longer be treated according to the study therapy. Patients of group B may get a HIPEC intervention without surgical cytoreduction if contraindication to the drugs applied can be excluded.

DETAILED DESCRIPTION:
The objective of the trial is to compare the treatment of patients with peritoneal metastasized gastric cancer including carcinoma of the AEG (Adenocarcinoma of the oesophago-gastric-junction) without evidence of other distant metastases treated with neoadjuvant chemotherapy followed by cytoreduction with intraperitoneal chemoperfusion (HIPEC) and postoperative chemotherapy (Group B) and patients treated with cytoreduction alone after neoadjuvant chemotherapy and postoperative chemotherapy (Group A).

Hypothesis of the trial is that surgical cytoreduction with intraperitoneal chemoperfusion (Group B) is superior to cytoreduction alone (Group A) in terms of overall survival.

The trial is designed as a prospective, randomized, open, multicenter and parallel group study.

ELIGIBILITY:
Inclusion Criteria:

* Histological proved diagnosis of peritoneal metastasized gastric cancer including carcinoma of the AEG No evidence of other distant metastases than peritoneal carcinomatosis with exception of Krukenberg Tumors
* Peritoneal Staging with laparoscopy (or explorative laparotomy) and estimation of Peritoneal Cancer Index (PCI) with the possibility of 80% tumor reduction at cytoreductive surgery
* Karnofsky Index 70% or better
* Written informed consent is obtained prior to commencement of trial treatment

Exclusion Criteria:

* Other than peritoneal metastasis of the gastric cancer incl. AEG and Krukenberg tumors
* Previous or concurrent malignancies, with the exception of adequately treated basal cell carcinoma of the skin or in situ carcinoma of the cervix
* Any previous chemotherapy or radiotherapy, and any investigational treatment for gastric cancer
* Active systemic infections
* Patients with known interstitial lung disease with New York Heart Association classification > 2
* Serious cardiac dysrhythmia or condition, New York Heart Association classification of III or IV, congestive cardiac failure
* cardiac arrhythmia
* Uncontrolled hypertension (diastolic blood pressure constantly >100 mm Hg, systolic blood pressure constantly > 180 mm Hg).
* Inadequate bone marrow function at the beginning of the trial, defined as platelet count less than <150 GPT/L or neutrophil granulocyte count less than <1.5 GPT/L
* cardiac function EF < 55%
* Inadequate renal function at the beginning of the trial, defined as GFR less than <60 ml/min
* Inadequate liver function at the beginning of the trial, defined as Bilirubin >1.5 times ULN
* Active vaccination within 6 weeks prior to randomisation
* Active hepatitis B or C infection
* Female patients who are pregnant or breast feeding
* Fertile female patients (defined as women with less than a 12-month elapse after the last menstruation) not using an acceptable form of contraception during the trial
* Missing of capacity to contract
* contraindication to the drugs which are used in the trial
* Participation in another therapeutic clinical trial
* Persons institutionalised due to regulatory actions ore by court order.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is overall survival | Death or 2.5 years
  Overall survival from randomisation up to end of study, follow up every 3 months till 2.5 years

SECONDARY OUTCOMES:
30 days complication-rate | 30 days postoperative
  30 days complication-rate. Complications are ranked from grade 0-5 according to CTCAE V4.0
time to progress | follow up every 3 months till 2.5 years end of study, 2.5 years
  time to progress of tumor, follow up every 3 months till 2.5 years
time to other distant metastases | end of study follow up every 3 months till 2.5 years
  time to other distant metastases follow up every 3 months till 2.5 years
quality of life | Every 6 months to 2,5 years
  quality of life (EORTC QLQ-30, STO 22). Every 6 months to 2,5 years

OTHER OUTCOMES:
frequency of toxicity and adverse events | every 3 weeks) and thereafter every 3 months up to 2.5 years end of study
  frequency of toxicity and adverse events, visit 1-11 (every 3 weeks) and thereafter every 3 months up to 2.5 years. AE is documented with the date of the begin and the end of the AE and the intensity according to CTCAE V4.0
frequency of necessary secondary surgical procedures and the length of hospitalisation | end of study, every 6 months up to 2.5 years
  frequency of necessary secondary surgical procedures and the length of hospitalisation every 6 months up to 2.5 years . The date of the begin and the end is daocumented as well as the reasons

CONTACTS AND LOCATIONS:
Overall Officials: Beate Rau, Prof., Study Director — Charite University, Berlin, Germany
Locations (1):
- Klinik für Allgemein-, Visceral-, Gefäß- und ThoraxchirurgieCharité Campus Mitte, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rau B, Lang H, Koenigsrainer A, Gockel I, Rau HG, Seeliger H, Lerchenmueller C, Reim D, Wahba R, Angele M, Heeg S, Keck T, Weimann A, Topp S, Piso P, Brandl A, Schuele S, Jo P, Pratschke J, Wegel S, Rehders A, Moosmann N, Gaedcke J, Heinemann V, Trips E, Loeffler M, Schlag PM, Thuss-Patience P. Effect of Hyperthermic Intraperitoneal Chemotherapy on Cytoreductive Surgery in Gastric Cancer With Synchronous Peritoneal Metastases: The Phase III GASTRIPEC-I Trial. J Clin Oncol. 2024 Jan 10;42(2):146-156. doi: 10.1200/JCO.22.02867. Epub 2023 Oct 31. PMID 37906724